CLINICAL TRIAL: NCT03242941
Title: AF Septal Pacing (Clinical Investigation Plan)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AF Septal Pacing
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Results first posted 2019-05-20 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Approximately 15 subjects with AF indicated for ablation of the pulmonary vein will be enrolled in the study. Participants will attend the Baseline visit and the Procedure visit. The baseline visit can be on the same day as the ablation procedure. Since it is an acute study, no follow-up visit will occur. The research procedure will be performed during an already scheduled ablation procedure. Subjects will be enrolled over a period of approximately 18 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persistent and Paroxtmal AF Patients (Experimental): Patients with either paroxymal or persistent AF already referred to the center for Pulmonary Vein Ablation will be stimulated delivering a novel dual-stage pacing protocol to terminate atrial fibrillation usinf a ring of electrodes positioned on the septum.
  Interventions: Procedure: Pulmonary vein ablation

INTERVENTIONS:
Procedure: Pulmonary vein ablation — After pulmonary vein isolation, during the routine waiting time of half an hour to confirm efficacy of the ablation, the septal catheter, already in place in right atrium, will be positioned on the interatrial septum. If the patient will not be in sinus rhythm, he/she will be externally cardioverted in order to determine pacing thresholds and impedances on all septal catheter electrodes. Next, atrial fibrillation will be induced by rapid atrial pacing.AF cycle length will be determined in the left atrial appendage, during 1 minute of atrial fibrillation using ablation catheter electrodes. Subsequently, a pacing scheme will be applied and capture on decapolar recording catheters, already in place for the standard ablation procedure will be assessed as well as AF termination.

SUMMARY:
The purpose of this non-randomized, non-controlled, acute, single-arm research study is to evaluate the feasibility to obtain a stable position of a ring of stimulation electrodes on the interatrial septum. The possibility to terminate atrial arrythmias will also be evaluated.

DETAILED DESCRIPTION:
The evidence of treating AF by pacing is limited, although these algorithms are of interest, since they appear to be safe and usually add little additional cost.

Using a computer model, a new dual-stage septal pacing has been developed.The proposed septal pacing algorithm could suppress AF reentries in a more robust way than classical single site rapid pacing. The feasibility of pacing both atria simultaneously from a single lead placed in the interatrial septum has been previously demonstrated clinically. The septal pacing concept has also been successfully tested in a computer model of AF and in a pig model . Experimental studies are now needed to determine whether similar termination mechanisms and efficacies can be observed in humans.

The purpose of this non-randomized, non-controlled, acute, single-arm research study is to evaluate the feasibility to obtain a stable position of a ring of stimulation electrodes on the interatrial septum

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to the center to undergo ablation of the pulmonary vein using radiofrequency (initial AF ablation, or redo procedure).
* In case of paroxysmal AF the right atrium should be dilated as indicated by > 29 ml mm2 or the left atrium should be dilated as indicated by > 34 ml mm2.
* Patient is willing and able to cooperate with the study procedure.
* Patient is willing to provide the Informed Consent for their participation in the study.

Exclusion Criteria:

* Patients under 18 years or over 80 years old.
* Women who are currently pregnant or have a positive pregnancy test.
* Patients with an implantable cardiac device.
* Patients who already underwent an AF septal ablation procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas V.A. Boersma, Principal Investigator — St. Antonius Hospital
Locations (3):
- Gottsegen György Országos Kardiológiai Intézet, Budapest, Hungary
- Netherlands (2):
  - Maastricht Universitair Medisch Centrum (MUMC), Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If the pulmonary vein ablation succeeded and the subject was in sinus rhythm the study procedure started from the electrode testing. Alternatively, if the subject was still in AF, the electrode testing was performed after either the application of the dual stage pacing algorithm or the cardioversion, when the sinus rhythm was established.
Groups:
- Persisten and Paroxymal AF Patients: Patients with either paroxymal or persistent AF already referred to the center for Pulmonary Vein Ablation will be stimulated delivering a novel dual-stage pacing protocol to terminate atrial fibrillation.
  Pulmonary vein ablation: After pulmonary vein isolation, during the routine waiting time of half an hour to confirm efficacy of the ablation, the septal catheter, already in place in right atrium, will be positioned on the interatrial septum. If the patient will not be in sinus rhythm, he/she will be externally cardioverted in order to determine pacing thresholds and impedances on all septal catheter electrodes. Next, atrial fibrillation will be induced by rapid atrial pacing.AF cycle length will be determined in the left atrial appendage, during 1 minute of atrial fibrillation using ablation catheter electrodes. Subsequently, a pacing scheme will be applied and capture on decapolar recording catheters will be assessed as well as AF termination.
Period: Overall Study
Arm/Group | Persisten and Paroxymal AF Patients
Started | 16
Completed | 14
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Paroxymal and Persistent AF Patients: Patients with either paroxymal or persistent AF already referred to the center for Pulmonary Vein Ablation will be stimulated delivering a novel dual-stage pacing protocol to terminate atrial fibrillation.
  Pulmonary vein ablation: After pulmonary vein isolation, during the routine waiting time of half an hour to confirm efficacy of the ablation, the septal catheter, already in place in right atrium, will be positioned on the interatrial septum. If the patient will not be in sinus rhythm, he/she will be externally cardioverted in order to determine pacing thresholds and impedances on all septal catheter electrodes. Next, atrial fibrillation will be induced by rapid atrial pacing.AF cycle length will be determined in the left atrial appendage, during 1 minute of atrial fibrillation using ablation catheter electrodes. Subsequently, a pacing scheme will be applied and capture on decapolar recording catheters will be assessed as well as AF termination.
Arm/Group | Paroxymal and Persistent AF Patients
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 182 (14)
Weight [Mean (Standard Deviation); unit: kg] | 92 (20)

OUTCOME MEASURES:

1. Primary Outcome: Number of Electrodes in a Stable Position
Description: To assess Pacing Site Stability, the number of interatrial septal pacing electrodes which are successfully placed in a stable position, will be counted. A stable position in this study is defined as a location where the pacing threshold will be < 10 mA at a pacing pulse width of 1 msec. Stable pacing further requires that no ventricular capture will be induced during atrial stimulation at twice the atrial capture threshold.
Time Frame: 30 minutes
Population: The maximum number of electrode pairs used and potentially stable
Measure: Count of Units; unit: Electrode pairs
Units Other Than Participants: Electrode pairs
Arm/Group | Paroxymal and Persistent AF Patients
Number analyzed (Participants) | 14
Number analyzed (Electrode pairs) | 60
Electrode pairs | 38

2. Secondary Outcome: Localized Atrial Capture
Description: To assess Localized Atrial Capture the following endpoints will be considered:
  - the number of AF episodes in which local capture is recorded during atrial septal stimulation in at least one of the electrode positions
Time Frame: 30 minutes
Population: Patient treated with the new pacing scheme algorithm
Measure: Count of Units; unit: Episodes
Units Other Than Participants: Episodes
Groups:
- Paroxymal or Persistent AF Patients: Patients with either paroxymal or persistent AF already referred to the center for Pulmonary Vein Ablation will be stimulated delivering a novel dual-stage pacing protocol to terminate atrial fibrillation.
  Pulmonary vein ablation: After pulmonary vein isolation, during the routine waiting time of half an hour to confirm efficacy of the ablation, the septal catheter, already in place in right atrium, will be positioned on the interatrial septum. If the patient will not be in sinus rhythm, he/she will be externally cardioverted in order to determine pacing thresholds and impedances on all septal catheter electrodes. Next, atrial fibrillation will be induced by rapid atrial pacing.AF cycle length will be determined in the left atrial appendage, during 1 minute of atrial fibrillation using ablation catheter electrodes. Subsequently, a pacing scheme will be applied and capture on decapolar recording catheters, already in place for the standard ablation procedure will be assessed as well
Arm/Group | Paroxymal or Persistent AF Patients
Number analyzed (Participants) | 14
Number analyzed (Episodes) | 14
Episodes | 8

3. Secondary Outcome: Termination of Atrial Tachyarrhythmia.
Description: Termination of atrial tachyarrhythmia.
Time Frame: 30 minutes
Population: Patients treated with the new dual stage pacing algorithm
Measure: Count of Units; unit: AF termination occurrence
Units Other Than Participants: AF termination occurrence
Arm/Group | Paroxymal or Persistent AF Patients
Number analyzed (Participants) | 14
Number analyzed (AF termination occurrence) | 14
AF termination occurrence | 3

ADVERSE EVENTS:
Time Frame: Since AF Septal Pacing is an acute study with no follow up and patient exit at the end of the procedure, only AE occurred during the procedure were recorded.
Description: Adverse Events were evaluated according to ISO 14155:2011
Arm/Group | Paroxymal and Persistent AF Patients
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxymal and Persistent AF Patients (N=14)
pericardial effusion (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT03242941/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03242941/SAP_001.pdf